CLINICAL TRIAL: NCT02307253
Title: EUS-guided Fine Needle Tissue Acquisition Using a Newly Developed Nitinol Ultra Flex 19 Gauge Needle for Transduodenal Lesions: a Multicenter Prospective Feasibility Study
Brief Title: EUS GUIDED Transduodenal Biopsy Using the 19G Flex
Acronym: NIFLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor of Surgery, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7427/13
Record Dates: First submitted 2014-11-19; First posted 2014-12-04 (Estimated); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-05

CONDITIONS: Abdominal Neoplasms
Keywords: EUS-guided biopsy, EUS-FNB
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with solid lesions (Experimental): Expect™19Flex needle (Boston Scientific Corp.,Natick,MA,USA)
  Interventions: Device: Expect™19Flex needle (Boston Scientific Corp.,Natick,MA,USA)

INTERVENTIONS:
Device: Expect™19Flex needle (Boston Scientific Corp.,Natick,MA,USA) — EUS-guided fine needle biopsy performed through the duodenum with the Expect™ 19 Flex needle

SUMMARY:
This study evaluates the feasibility, safety and accuracy of a 19 gauge (19G) needle in nitinol in the performance of endoscopic ultrasound (EUS) guided transduodenal biopsy for the acquisition of samples for histologic analysis. Patients with lesions that can be approached only from the duodenum will be prospectively enrolled.

DETAILED DESCRIPTION:
A 19 gauge needle in nitinol (Flex needle) has been recently become available for EUS guided procedure.

The use of nitinol should guarantee a better needle flexibility with a theoretical advantage on the use of this needle for lesions that need to be sampled through the duodenum. Moreover, samples for histologic examination seems to be easy to interpret than cytologic ones allowing evaluate of the overall architecture of the tissue, better performance of immunohistochemical staining, and may be of additional value to perform tissue profiling that in the future will be very important to guide individualized therapies

The existing data on the performance of the Flex needle for EUS-guided transduodenal biopsy are coming form a single study performed in one single center. Thus, the reproducibility of these results is unknown and multicenter prospective studies are warranted to answer this important question.

ELIGIBILITY:
Inclusion Criteria:

A. Age greater than 18 and less than 90. B. Presence of a solid lesion of the gastrointestinal tract adjacent to the duodenum with no previous tissue diagnosis.

C. Absence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma.

D. Informed consent is obtained.

Exclusion Criteria:

A. Presence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma.

B. Altered anatomy of the upper gastrointestinal tract due to surgery of the esophagus, stomach and duodenum.

C. They are unable to understand and/or read the consent form.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Costamagna, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (6):
- Indiana Univerisity Health Medical Center, Indianapolis, Indiana, United States
- Clinique du Trocadero, Paris, France
- Italy (3):
  - AUSL Bologna Bellaria-Maggiore Hospital, Bologna
  - ISMETT UPMC Italy, Palermo
  - Digestive Endoscopy Unit, Universita' Cattolica del Sacro Cuore, Rome
- Teikyo University Mizonokuchi Hospital, Departement of Gastroenterology, Kawasaki, Kanagawa, Japan

REFERENCES:
- [Result] Varadarajulu S, Bang JY, Hebert-Magee S. Assessment of the technical performance of the flexible 19-gauge EUS-FNA needle. Gastrointest Endosc. 2012 Aug;76(2):336-43. doi: 10.1016/j.gie.2012.04.455. PMID 22817786

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: consecutive patients with solid lesions who needed to undergo EUS for tissue sampling that had to be performed through the duodenum, such as for deep head/uncinate pancreatic masses, periduodenal lymph nodes, duodenal subepithelial lesions, aortocaval nodes, hilar tumors, right-sided liver lesions, right kidney lesions, right adrenal gland lesions, or periduodenal abdominal masses, were enrolled in the present study.
Period: Overall Study
Arm/Group | Patients With Solid Lesions
Started | 246
Completed | 246
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Solid Lesions: all consecutive patients with solid lesions who needed to undergo EUS for tissue sampling that had to be performed through the duodenum, such as for deep head/uncinate pancreatic masses, periduodenal lymph nodes, duodenal subepithelial lesions, aortocaval nodes, hilar tumors, right-sided liver lesions, right kidney lesions, right adrenal gland lesions, or periduodenal abdominal masses, were enrolled in the present study.
  Selection criteria All adults (>18 years of age) referred for EUS-FNA of solid lesions adjacent to or located in the wall of the duodenum with no previous tissue diagnosis were considered eligible. In the presence of a cystic component, the solid part of the lesion should have been more than 75% of the total. Patients with uncorrectable coagulopathy as defined by abnormal prothrombin time or partial thromboplastin time that did not normalize after administration of fresh frozen plasma, with altered anatomy of the upper GI tract due to surgery of the esophagus, stomach, and duodenum and those unable to understand and/or read the consent form were excluded from the current study.
Arm/Group | Patients With Solid Lesions
Number analyzed (Participants) | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 144
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
  Japan | 25
  Italy | 152
  France | 39

OUTCOME MEASURES:

1. Primary Outcome: Capability of Performing EUS-FNTA Through the Duodenum by Placing the Target Lesion in the Proper Position With Insertion of the Needle Into the Lesion
Description: Number of patients in which it was possible to place the needle within the target lesion by a transduodenal route divided by the total number of enrolled patients.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Solid Lesions
Number analyzed (Participants) | 246
Participants | 228

2. Secondary Outcome: Number of Complications Divided Per Total Number of Enrolled Patients
Description: rate of complications, divided in procedural complication (perforation, bleeding) occurring during the procedure and late complications (delayed bleeding, infection) occurring during the post-procedural observational period
Time Frame: intraoperative and within 3 days after the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Solid Lesions
Number analyzed (Participants) | 246
Participants | 6

3. Secondary Outcome: Number of Histological Samples Judged Adequate Divided by the Total Number of Patients
Description: percentage of patients in whom a histologically interpretable specimen will be retrieved
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Solid Lesions
Number analyzed (Participants) | 246
Participants | 189

4. Secondary Outcome: Number of Correct Diagnosis Divided by the Total Number of Patients
Description: rate of correct diagnosis obtained through analysis of the tissue samples acquired with EUS fine needle biopsy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Solid Lesions
Number analyzed (Participants) | 246
Participants | 181

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients With Solid Lesions
Serious Adverse Events (participants affected / at risk) | 6/246
Other Adverse Events (participants affected / at risk) | 0/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Solid Lesions (N=246)
Bleeding (Gastrointestinal disorders) | 2 (2)
acute pancreatitis (Hepatobiliary disorders) | 2 (2)
duodenal perforation (Gastrointestinal disorders) | 1 (1)
duodenal hematoma (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No